CLINICAL TRIAL: NCT04185896
Title: Perinatal Mental Health Care in Switzerland: Unraveling the Perspectives of Affected Women and Health Professionals
Brief Title: Perinatal Mental Health Care in Switzerland
Acronym: MADRE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bern University of Applied Sciences (Other)
Collaborators: University of Bern (Other)
Responsible Party: Principal Investigator, Anke Berger, Project leader, Bern University of Applied Sciences
Other Study IDs: 2218-2018
Record Dates: First submitted 2019-11-19; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Mental Disorder; Perinatal; Depression; Anxiety Disorders; Panic Disorder; Post Traumatic Stress Disorder; Adaptation Reaction; Behavior Disorders; Substance Abuse; Psychosis; Health Care Seeking Behavior; Health Care Utilization; Health Care Acceptability
Keywords: Social stigma; Access to care; Facilitators; Barriers
MeSH Terms: conditions — Mental Disorders; Depression; Anxiety Disorders; Panic Disorder; Stress Disorders, Post-Traumatic; Substance-Related Disorders; Psychotic Disorders; Patient Acceptance of Health Care; Social Stigma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This qualitative study with quantitative elements examines the health care provided to women who suffered from mental disorder during pregnancy and / or in the first year after birth (i.e. during the perinatal phase). Investigators will perform individual interviews with former PMD patients, and health and social care professionals to gain insights into current health care for PMD patients.

DETAILED DESCRIPTION:
Background: Perinatal mental disorders (PMD) are highly prevalent (up to 20%), and patients use mental health care at high rates (Berger et al 2018). It is not known if the health care for PMD patients meets the needs of the patients.

Aim: The Investigators will identify factors that promote or hinder service provision and access to care, for a range of relevant PMD. The investigation will cover the user and provider perspectives.

Methods: The qualitative study consists of two complementary parts to assess user and provider perspectives. In part 1 the Investigators will conduct individual semi-structured interviews with 24 women who have had PMD. The sample will comprise of 4 clusters of relevant ICD-10 F-diagnoses, covering a wide range of mental disorders. The sample will also comprise of participants who received or did not receive mental health care before the last pregnancy. In part 2, the Investigators perform 3 focus groups (with 6-8 participants per group) with health and social care professionals, and a health-insurance delegate, to collect their experiences and perspectives on perinatal health care for PMD patients. The Investigators are guided for data collection and analysis by Levesque's et al (2013) conceptual model on access to health care.

Expected results: The study will identify barriers and facilitators for health care access (user perspective) and provision (provider perspective). The study will generate the evidence base needed to develop integrated, coordinated, patient- and family-centered care for patients with various types of PMD.

ELIGIBILITY:
Sample 1: patients with former PMD

Inclusion criteria:

1. PMD within the past 24 months before the interview,
2. Recovered from acute PMD and stable for at least 12 months before the interview;
3. Able to share experiences;
4. More than 18 years old
5. Speak and understand German
6. At least 1 diagnosis in the last perinatal phase out of 4 groups of psychiatric disorders (ICD-10 Chapter V, F00-F99):

   1. Mood (affective) disorders (F30-F39); Anxiety disorders (F41); Reaction to severe stress, and adjustment disorders (F43); and Obsessive-compulsive disorder (F42);
   2. Disorders of adult personality and behavior (F60-F69; especially F60.3 Emotionally unstable personality disorder);
   3. Mental and behavioral disorders due to psychoactive substance use (F10-F19; excluding tobacco (F17) if it is the sole F-diagnosis of the patient);
   4. Psychosis (F20-F29 Schizophrenia, schizotypal and delusional disorders).

Exclusion criterion: Current pregnancy

Sample 2: Professional health and social care providers

Inclusion criteria:

1. Professional experience of at least two years,
2. Have cared for at least 2 PMD patients the year before the focus group, a
3. Speak and understand German.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population 1: 24 former PMD patients, by 4 groups of F-diagnoses (ICD-10) and 2 groups (yes or no) of pre-existent mental disorders.
  Population 2: 18-24 professional health care and social care providers, who are experienced in service provision for PMD patients and are
  * Nurses
  * Midwives
  * Gynecologists
  * Medical primary care providers
  * Pediatricians
  * Neonatologists
  * Psychiatrists
  * Psychologists
  * Social care providers (community service)
  * Expert from a health insurance
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-02-29 (Estimated); Study Completion 2020-02-29 (Estimated)

PRIMARY OUTCOMES:
Narratives of barriers to perinatal mental health care use | perinatal phase, i.e. pregnancy and first year after birth
  Narratives of access-inhibiting factors, in semi-structured individual interviews with former PMD patients
Narratives of mentions of facilitators of perinatal mental health care use | Perinatal phase, i.e. pregnancy and first year after birth
  Narratives of access-promoting factors, in semi-structured individual interviews with former PMD patients
Narratives of mentions of barriers to perinatal mental health care provision | Perinatal phase, i.e. pregnancy and first year after birth
  Narratives of provision-inhibiting factors, in focus group interviews with health and social care providers
Narratives of mentions of facilitators of perinatal mental health care provision | Perinatal phase, i.e. pregnancy and first year after birth
  Narratives of provision-promoting factors, in focus group interviews with health and social care providers

SECONDARY OUTCOMES:
Sociodemographic data of participating affected PMD patients | 2019-2020
  Sociodemographic data of participating affected PMD patients
Sociodemographic data of participating health care professionals | 2019-2020
  Sociodemographic data of participating health care professionals

CONTACTS AND LOCATIONS:
Locations (1):
- Anke Berger, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
The Ethics Committee does not allow sharing of patients' data. The Ethics Committee allows and the Investigators are willing to share the data collected from health and social care professionals upon publication of the study.

REFERENCES:
- [Background] Berger A, Bachmann N, Signorell A, Erdin R, Oelhafen S, Reich O, Cignacco E. Perinatal mental disorders in Switzerland: prevalence estimates and use of mental-health services. Swiss Med Wkly. 2017 Mar 7;147:w14417. doi: 10.4414/smw.2017.14417. eCollection 2017. PMID 28322424
- [Derived] Berger A, Schenk K, Ging A, Walther S, Cignacco E. Perinatal mental health care from the user and provider perspective: protocol for a qualitative study in Switzerland. Reprod Health. 2020 Feb 17;17(1):26. doi: 10.1186/s12978-020-0882-7. PMID 32066475